CLINICAL TRIAL: NCT01437332
Title: Molecular Mediators of Nerve Injury Signaling
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0356-11-RMB
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes; Nerve Injury; Chronic Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Diabetes
- Nerve injury
- Other

SUMMARY:
Specific proteins and other signaling molecules are increased and decreased following nerve injury. Some of these are important in producing pain or explaining why pain persists after traumatic nerve injuries or in disease states such as diabetes. In this study, the investigators hypothesize that it is possible to detect changes in specific signaling molecules and that these will provide insights into novel treatment strategies. The patients to be included are those who are undergoing the removal of tissue during surgery. The tissues that would otherwise be discarded will be included in the study as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery where tissue removal is anticipated

Exclusion Criteria:

* age younger than 18

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical procedures at Rambam Health Care Campus wherein the surgeon and PI determine appropriateness for study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-09 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Ebenezer GJ, McArthur JC, Thomas D, Murinson B, Hauer P, Polydefkis M, Griffin JW. Denervation of skin in neuropathies: the sequence of axonal and Schwann cell changes in skin biopsies. Brain. 2007 Oct;130(Pt 10):2703-14. doi: 10.1093/brain/awm199. PMID 17898011